CLINICAL TRIAL: NCT03284424
Title: A Phase 2, Open-Label, Single Arm Study to Evaluate the Safety and Efficacy of Pembrolizumab in Participants With Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (R/M cSCC)
Brief Title: Study of Pembrolizumab (MK-3475) in Adults With Recurrent/Metastatic Cutaneous Squamous Cell Carcinoma (cSCC) or Locally Advanced Unresectable cSCC (MK-3475-629/KEYNOTE-629)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-629; MK-3475-629 (Other: Merck); KEYNOTE-629 (Other: Merck); 2017-000594-37 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: Squamous Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Squamous Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- R/M cSCC cohort (Experimental): Participants with R/M cSCC receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab
- LA cSCC cohort (Experimental): Participants with LA cSCC receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pembrolizumab (MK-3475) in adult participants with recurrent or metastatic(R/M) cutaneous Squamous Cell Carcinoma (cSCC) or locally advanced (LA) unresectable cSCC that is not amenable to surgery and/or radiation and/or systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* R/M cSCC cohort only:
* Has cSCC that is either metastatic defined as disseminated disease, and/or unresectable disease that is not curable by surgery or radiation.
* Has histologically-confirmed cSCC as the primary site of malignancy (metastatic skin involvement from another primary cancer or from an unknown primary cancer is not permitted).
* LA cSCC cohort only:
* Must be ineligible for surgical resection.
* Participants who received prior radiation therapy (RT) to index site or must be deemed to be not eligible for RT.
* Participants who received prior systemic therapy for curative intent are eligible regardless of regimen.
* R/M cSCC cohort only:
* Has metastatic disease defined as disseminated disease distant to the initial/primary site of diagnosis, and/or must have locally recurrent disease that has been previously treated (with either surgery or radiotherapy), and is not amenable to either curative surgery or radiotherapy.
* Has measurable disease based on RECIST 1.1 as assessed by the central imaging vendor.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 10 days prior to the start of study treatment.
* Has adequate organ function.
* Has a tissue sample adequate for programmed death-ligand 1 (PD-L1) testing as determined by central laboratory testing prior to study allocation.
* Has a life expectancy >3 months.
* Female participants of childbearing potential must agree to use an adequate method of contraception during the study treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

* Has cSCC that can be cured with surgical resection, radiotherapy, or with a combination of surgery and radiotherapy.
* Has any other histologic type of skin cancer other than invasive squamous cell carcinoma as the primary disease under study, e.g. basal cell carcinoma that has not been definitively treated with surgery or radiation, Bowen's disease, Merkel cell carcinoma (MCC), melanoma.
* Has had any prior allogeneic solid organ or bone marrow transplantation.
* Has received prior therapy with an anti-programmed death protein-1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g. cytotoxic T-lymphocyte associated protein 4 [CTLA-4], Tumor necrosis factor receptor superfamily, member 4 [OX-40], tumor necrosis factor receptor superfamily member 9 [CD137]).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study allocation.

(Notes: Participants must have recovered from all AEs due to previously administered therapies to ≤ Grade 1 or baseline. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.)

* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (e.g. with use of disease-modifying agents, anticoagulants, corticosteroids or immunosuppressive drugs).
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (59):
- United States (14):
  - Moores UC San Diego Cancer Center ( Site 0352), La Jolla, California
  - Stanford University Medical Center ( Site 0366), Palo Alto, California
  - St. Joseph Heritage Healthcare ( Site 0350), Santa Rosa, California
  - Yale University ( Site 0365), New Haven, Connecticut
  - Lombardi Comprehensive Cancer Center ( Site 0360), Washington D.C., District of Columbia
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 0353), Indianapolis, Indiana
  - University of Kansas Cancer Center ( Site 0361), Westwood, Kansas
  - Massachusetts General Hospital ( Site 0362), Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada ( Site 8001), Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack University Med Ctr ( Site 0367), Hackensack, New Jersey
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0364), Tulsa, Oklahoma
  - Fox Chase Cancer Center ( Site 0351), Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 0356), Sioux Falls, South Dakota
  - Texas Oncology PA ( Site 8000), Dallas, Texas
- Australia (6):
  - Orange Health Services ( Site 0406), Orange, New South Wales
  - Southern Medical Day Care Centre ( Site 0408), Wollongong, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0407), Herston, Queensland
  - Princess Alexandra Hospital ( Site 0405), Woolloongabba, Queensland
  - The Townsville Hospital ( Site 0404), Douglas
  - Lismore Base Hospital ( Site 0402), Lismore
- Canada (5):
  - Dr. Leon Richard Oncology Centre ( Site 0100), Moncton, New Brunswick
  - The Ottawa Hospital Cancer Centre ( Site 0101), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0105), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0102), Toronto, Ontario
  - Jewish General Hospital ( Site 0103), Montreal, Quebec
- France (10):
  - IUCT - Oncopole ( Site 0604), Toulouse, Cedex 9
  - Hopital Avicenne ( Site 0609), Bobigny
  - CHRU Lille - Hopital Claude Huriez ( Site 0605), Lille
  - CHU Limoges CHU Dupuytren ( Site 0608), Limoges
  - Hopital La Timone ( Site 0603), Marseille
  - Hopital Archet 3 ( Site 0607), Nice
  - Hopital Saint-Louis ( Site 0601), Paris
  - CH Lyon Sud Hospices Civils de Lyon ( Site 0600), Pierre-Bénite
  - CHU Reims - Hopital Robert Debre ( Site 0610), Reims
  - Institut Gustave Roussy (IGR) ( Site 0602), Villejuif
- Germany (5):
  - Universitaetsklinikum Essen ( Site 0650), Essen
  - Medizinische Hochschule Hannover ( Site 0652), Hanover
  - Universitaets-Hautklinik Kiel ( Site 0656), Kiel
  - Universitaetsklinikum Mannheim GmbH ( Site 0654), Mannheim
  - Universitatsklinikum Tübingen ( Site 0651), Tübingen
- Israel (4):
  - Rambam Health Care Campus ( Site 0950), Haifa
  - Rabin Medical Center ( Site 0952), Petah Tikva
  - Sheba Medical Center ( Site 0953), Ramat Gan
  - Sourasky Medical Center. ( Site 0951), Tel Aviv
- Mexico (4):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0301), Guadalajara, Jalisco
  - Hospital y Clinica OCA SA de CV/Monterrey International ResearchCenter ( Site 0306), Monterrey, Nuevo León
  - Centro Estatal de Cancerologia de Chihuahua ( Site 0308), Chihuahua City
  - Grupo Medico Camino SC ( Site 0300), Mexico City
- Norway (2):
  - Haukeland Universitetssykehus ( Site 0902), Bergen
  - Oslo Universitetssykehus Radiumhospitalet ( Site 0901), Oslo
- Spain (5):
  - Hospital Duran i Reinals ICO de Hospitalet ( Site 0751), Hospitalet Del Llobregat, Barcelona
  - Hospital Vall D Hebron ( Site 0750), Barcelona
  - Hospital Clinic i Provincial Barcelona ( Site 0754), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 0753), Madrid
  - Hospital General de Valencia ( Site 0752), Valencia
- United Kingdom (4):
  - The Clatterbridge Cancer Centre NHS Foundation Trust ( Site 0803), Bebington, Wirral
  - University College Hospital NHS Foundation Trust ( Site 0801), London
  - Royal Marsden NHS Foundation Trust ( Site 0800), London
  - Royal Cornwall Hospitals NHS Trust ( Site 0804), Truro

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Grob JJ, Gonzalez R, Basset-Seguin N, Vornicova O, Schachter J, Joshi A, Meyer N, Grange F, Piulats JM, Bauman JR, Zhang P, Gumuscu B, Swaby RF, Hughes BGM. Pembrolizumab Monotherapy for Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma: A Single-Arm Phase II Trial (KEYNOTE-629). J Clin Oncol. 2020 Sep 1;38(25):2916-2925. doi: 10.1200/JCO.19.03054. Epub 2020 Jul 16. PMID 32673170
- [Derived] Bratland A, Munoz-Couselo E, Mortier L, Roshdy O, Gonzalez R, Schachter J, Arance AM, Grange F, Meyer N, Joshi AJ, Billan S, Hughes BGM, Grob JJ, Ramakrishnan K, Ge J, Gumuscu B, Swaby RF, Gutzmer R. Health-Related Quality of Life with Pembrolizumab in Patients with Locally Advanced or Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma: KEYNOTE-629. Dermatol Ther (Heidelb). 2023 Dec;13(12):3165-3180. doi: 10.1007/s13555-023-01059-y. Epub 2023 Nov 9. PMID 37943491
- [Derived] Hughes BGM, Mendoza RG, Basset-Seguin N, Vornicova O, Schachter J, Joshi A, Meyer N, Grange F, Piulats JM, Bauman JR, Chirovsky D, Zhang P, Gumuscu B, Swaby RF, Grob JJ. Health-Related Quality of Life of Patients with Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma Treated with Pembrolizumab in KEYNOTE-629. Dermatol Ther (Heidelb). 2021 Oct;11(5):1777-1790. doi: 10.1007/s13555-021-00598-6. Epub 2021 Sep 23. PMID 34558040
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 2 cohorts in this study and each cohort received the same dose/treatment regimen. Participant flow, baseline characteristics, and outcome measures are presented by cohort. Adverse events were pre-specified to be reported as a single group by intervention for first and second course pembrolizumab.
Groups:
- Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (cSCC) Cohort: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 doses (approximately 24 months). Eligible participants who stopped the initial course of pembrolizumab but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Locally Advanced Unresectable cSCC Cohort: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 doses (approximately 24 months). Eligible participants who stopped the initial course of pembrolizumab but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Period: Overall Study
Arm/Group | Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (cSCC) Cohort | Locally Advanced Unresectable cSCC Cohort
Started | 105 | 54
Participants That Received a Second Course of Pembrolizumab | 2 | 1
Completed | 0 | 0
Not Completed | 105 | 54
Not completed — Death | 70 | 24
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Sponsor's decision | 27 | 22

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (cSCC) Cohort | Locally Advanced Unresectable cSCC Cohort | Total
Number analyzed (Participants) | 105 | 54 | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (14.3) | 73.7 (12.4) | 71.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 40
  Male | 80 | 39 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 2 | 15
  Not Hispanic or Latino | 57 | 40 | 97
  Unknown or Not Reported | 35 | 12 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 68 | 40 | 108
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 32 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who have best response of Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). ORR per RECIST 1.1 as assessed by blinded independent central review (BICR) is presented.
Time Frame: Up to approximately 32 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Recurrent or Metastatic Cutaneous cSCC Cohort; Locally Advanced Unresectable cSCC Cohort: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 doses (approximately 24 months).
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Percentage of participants | 35.2 [26.2 to 45.2] | 51.9 [37.8 to 65.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed CR or PR per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. The DOR per RECIST 1.1 as assessed by BICR is presented for all participants who experienced a confirmed CR or PR.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had confirmed complete response or partial response.
Measure: Median (Full Range); unit: Months
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 37 | 28
Months | 1.6 [1.2 to 24.7] | 2.7 [1.1 to 12.3]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who have a CR or PR or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease). The DCR per RECIST 1.1 as assessed by BICR is presented.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Percentage of participants | 52.4 [42.4 to 62.2] | 64.8 [50.6 to 77.3]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment to the first documented PD or death due to any cause, whichever occurred first. PFS per RECIST 1.1 as assessed by BICR is presented.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Months | 5.7 [3.1 to 8.5] | 14.4 [5.5 to 43.6]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment to death due to any cause. The OS for all participants is presented.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Months | 23.8 [13.4 to 30.9] | NA [33.3 to NA] — NA= Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

6. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Participants | 102 | 51

7. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AE
Description: An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 56 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent or Metastatic Cutaneous cSCC Cohort | Locally Advanced Unresectable cSCC Cohort
Number analyzed (Participants) | 105 | 54
Participants | 20 | 11

ADVERSE EVENTS:
Time Frame: Up to approximately 56 months
Description: The analysis population for AEs included all participants who received ≥1 dose of study treatment. Adverse Events were pre-specified to be reported as a single group by intervention for first course and second course. Per protocol, disease progression was not considered an AE unless considered related to study treatment. Therefore, MedDRA preferred terms "neoplasm progression (NP)", "malignant NP" and "disease progression" not related to study treatment are excluded.
Groups:
- Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC First Course: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 doses (approximately 24 months).
- Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC Second Course: Eligible participants who stopped the initial course of pembrolizumab but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Arm/Group | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC First Course | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC Second Course
All-Cause Mortality (participants affected / at risk) | 97/159 | 1/3
Serious Adverse Events (participants affected / at risk) | 87/159 | 2/3
Other Adverse Events (participants affected / at risk) | 139/159 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC First Course (N=159) | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Infestation (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (19) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC First Course (N=159) | Recurrent or Metastatic Cutaneous and Locally Advanced Unresectable cSCC Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 18 (26) | 0 (0)
Hypothyroidism (Endocrine disorders) | 14 (16) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 40 (47) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 31 (38) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (29) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (22) | 0 (0)
Asthenia (General disorders) | 35 (44) | 1 (1)
Chest pain (General disorders) | 8 (8) | 0 (0)
Fatigue (General disorders) | 35 (39) | 0 (0)
Oedema peripheral (General disorders) | 17 (21) | 0 (0)
Pyrexia (General disorders) | 14 (17) | 0 (0)
Bronchitis (Infections and infestations) | 8 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (10) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (13) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (1)
Blood creatinine increased (Investigations) | 8 (8) | 0 (0)
Blood phosphorus decreased (Investigations) | 2 (2) | 1 (1)
Blood urea increased (Investigations) | 2 (2) | 1 (2)
Protein total decreased (Investigations) | 1 (7) | 1 (3)
Weight decreased (Investigations) | 18 (19) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 25 (27) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (26) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (29) | 0 (0)
Dizziness (Nervous system disorders) | 11 (12) | 0 (0)
Headache (Nervous system disorders) | 18 (20) | 0 (0)
Paraesthesia (Nervous system disorders) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (10) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 9 (15) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (45) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 25 (34) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 10 (19) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03284424/Prot_SAP_001.pdf